CLINICAL TRIAL: NCT05367570
Title: Move, Sit, Sleep, Repeat: Exploring 24-hour Movement Behaviors Among Normal Weight, Overweight and Obese Adults and the Power of Co-created Interventions
Brief Title: 24-hour Movement Behaviors Among Normal Weight, Overweight and Obese Adults
Acronym: OwOb_24hmb
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0013
Record Dates: First submitted 2022-04-27; First posted 2022-05-10 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Overweight and Obesity
Keywords: physical activity; sedentary behavior; sleep; 24-hour movement behaviors
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood sample will be collected in order to analyze HbA1c, Cholesterol, glucose, triglycerides
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal weight group: The first work package of this study is cross-sectional. The investigators will investigate the 24-hour movement behaviors, cardiometabolic parameters and some personal and environmental correlates.
  Interventions: Behavioral: Cross-sectional observational study
- Overweight/obesity group: The first work package of this study is cross-sectional The investigators will investigate the 24-hour movement behaviors, cardiometabolic parameters and some personal and environmental correlates.
  Interventions: Behavioral: Cross-sectional observational study

INTERVENTIONS:
Behavioral: Cross-sectional observational study — The first work package of this project is an explanatory cross-sectional study with no intervention.

SUMMARY:
The prevalence of adults with overweight (50%) and obesity (15%) reached high number in Belgium. Important lifestyle behaviors, i.e. sleep, sedentary time (SB), and physical activity (PA) subdivided into light physical activity (LPA) and moderate to vigorous physical activity (MVPA), have shown an impact on overweight and obesity characteristics (e.g. adiposity). However, these behaviors have often been investigated separately. Therefore, a recent shift in research emphasizes the importance of considering these behaviors as part of a 24-hour day.

Since these adults can benefit from an optimal 24-hour composition as part of a healthy lifestyle, it may be interesting to investigate the 24-hour movement composition among these adults. In addition, exploring different personal determinants, environmental determinants, and cardiometabolic markers will provide meaningful insights in developing an intervention.

ELIGIBILITY:
Inclusion criteria OwOb group

* Adults aged 25-64 years
* Active on the job market for at least 50 percent
* BMI ≥25kg/m² and Waist Circumference C ≥94cm for men and ≥80 cm for women

Inclusion criteria Nw participants

* Adults aged 25-64 years
* Active on the job market for at least 50 percent
* BMI <25kg/m² and Waist Circumference <94cm for men and <80 cm for women

Exclusion criteria Nw, Ow, Ob patients

* Retirement and early retirement
* Unemployment
* Working for less than 50 percent
* Working in night shifts
* Physical (e.g. amputations, paralysis, recovering from stroke, osteoarthritis), cognitive (e.g. dementia, psychological disorders) and major medical (e.g. Chronic respiratory diseases, heart failure, cardiovascular diseases) conditions that obstruct daily functioning
* Taking diabetes related medication
* Active treatment for cancer
* Pregnancy
* Breastfeeding
* Pregnancy <1 year ago
* Currently involved in study specific weight loss interventions
* Waitlist for weight loss surgery
* Weight loss surgery <1 year ago
* Taking medication which affects your body weight (e.g. thyroid medication, psychotropic medication)
* Thyroid problems which affects your body weight
* Hospitalized

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: One hundred seventy-two adults will be distributed into a Nw group and an OwOb group. Based on the Health Survey (2018), the general Belgian population has a prevalence of 50 percent OwOb adults. Therefore the distribution in this cross-sectional study will follow these percentages: 50 percent Nw adults (n=86) and 50 percent OwOb adults (n=86). Based on the Health Survey (2018), the group of OwOb adults can be divided into 35 percent Ow adults and 15 percent Ob adults. This represents itself in the inclusion of 60 adults (35%) with overweight and 26 adults (15%) with obesity. Adults of the Nw group will be matched with the OwOb group based on sex and age.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
24-hour movement behaviors | Through study completion, an average of 6 months to 1 year
  During their visit to Ghent University hospital, participants will receive a 'wGT3X-BT' 'ActiGraph accelerometer that will objectively measure their 24-hour movement behaviors (PA, SB, and sleep). The participants will wear the accelerometer for seven consecutive days. Additionally, this accelerometer data will be supplemented with a diary to validate sleep time and (non)wear time.

SECONDARY OUTCOMES:
Demographics | Through study completion, an average of 6 months to 1 year
  The following demographics will be questioned: age, sex, marital status, family situation, living environment, ethnicity, smoking, educational level, profession, net family income, and medication intake, PA participation, dietary interventions
Dietary factors | Through study completion, an average of 6 months to 1 year
  A Food Frequency Questionnaire will collect dietary information. This questionnaire is based on the Flemish food-based dietary guidelines for adults. This questionnaire can make a distinction between following a healthy plant based diet and unhealthy plant based diet.
Quality of Life (QoL) | Through study completion, an average of 6 months to 1 year
  The Health related quality of life scale 'Short Form Health Survey' (SF-12) is classified into 8domains: physical functioning, role-physical, bodily pail, general health, energy/fatigue, social functioning, role-emotional, mental health. Scale is between 0 and 100 where a higher score reflects a better QoL.
Depression | Through study completion, an average of 6 months to 1 year
  The Beck Depression Inventory will be used to screen for depression among this target group. It is one of the most widely used depression instruments. It measures both the intensity of depression as well as a screening for depression in Nw and OwOb adults. The Scale is between 0 an 63 where a higher score reflects a higher susceptibility of depression.
Behavioral factors | Through study completion, an average of 6 months to 1 year
  The following behaviors will be questioned: autonomous motivation, attitude, self-efficacy, subjective norm, internal control (i.e. habits, routines, skills), and external control (i.e. perceived barriers, real barriers). These questions are part a self-developped questionnaire which is currently tested for reliability. The scores will be calculated based on the cumulative percentage of the group. A higher score reflects a higher score on the specific behavioral construct.
Environmental factor | Through study completion, an average of 6 months to 1 year
  The environmental factors are divided into socio-environmental factors and physical environmental factors. Socio-environmental factors are social support and modeling. Physical environmental factors are walkability, neighborhood, work environment, sleep environment, and electronic devices at home. These questions are part a self-developped questionnaire which is currently tested for reliability. The scores will be calculated based on the cumulative percentage of the group. A higher score reflects a higher score on the specific environmental construct.
HbA1c | Through study completion, an average of 6 months to 1 year
  Blood parameters will be collected by a study nurse. This blood sample will be collected in a EDTA tube and will be analyzed by the clinical lab of Ghent university Hospital.
Glucose | Through study completion, an average of 6 months to 1 year
  Blood parameters will be collected by a study nurse. This blood sample will be collected in a Serum tube and will be analyzed by the clinical lab of Ghent university Hospital.
Triglycerides | Through study completion, an average of 6 months to 1 year
  Blood parameters will be collected by a study nurse. This blood sample will be collected in a Serum tube and will be analyzed by the clinical lab of Ghent university Hospital.
Cholesterol (total, HDL, LDL) | Through study completion, an average of 6 months to 1 year
  Blood parameters will be collected by a study nurse. This blood sample will be collected in a Serum tube and will be analyzed by the clinical lab of Ghent university Hospital.
Body mass index | Through study completion, an average of 6 months to 1 year
  BMI will be calculated by measuring weight (Seca 861) and height (Seca 213). The weight and height will be used in this formula: BMI (kg/m²)= (weight in kg)/(height in m)².
Waist circumference | Through study completion, an average of 6 months to 1 year
  The waist circumference will be measured with a measuring tape (Seca 201).
waist to hip ratio (WHR) | Through study completion, an average of 6 months to 1 year
  The hip circumference will be measured with a measuring tape (Seca 201).Both waist and hip circumferences will be used to calculate WHR= (waist circumference in cm)/ (hip circumference in cm)
body fat percentage | Through study completion, an average of 6 months to 1 year
  The body fat percentage will measured by 'Tanita SC-240MA'
blood pressure | Through study completion, an average of 6 months to 1 year
  Blood pressure will be measured twice (interval of one minute) with an automatic OMRON M6 Comfort device after 10 minutes of rest
Advanced Glycation Endproducts (AGE's) | Through study completion, an average of 6 months to 1 year
  AGE's are interesting to explore as predictors in developing several comorbidities (e.g. cardiovascular diseases, microvascular complications). They will be measured with an AGE-reader, which is a quick and non-invasive device
Obstructive sleep apnea (OSA's) risk | Through study completion, an average of 6 months to 1 year
  To measure OSA's risk, I will measure the participants' neck circumference by a measuring tape (Seca 201) and ask questions based on the STOP-BANG questionnaire. Scale ranges between 0 and 8. A higher score reflects a higher risk for OSA.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Lapauw, Professor, Principal Investigator — Ghent University Hospital - endocrinologist; Marieke De Craemer, Professor, Principal Investigator — University Ghent
Locations (1):
- Ghent University Hospital, Dept. of Endocrinoly, Ghent, East-Flanders, Belgium